CLINICAL TRIAL: NCT01488526
Title: Tenofovir Disoproxil Fumarate in Late Pregnancy to Prevent Vertical Transmission of Hepatitis B Virus in Highly Viremic Mothers
Brief Title: Tenofovir in Late Pregnancy to Prevent Vertical Transmission of Hepatitis B Virus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New Discovery LLC (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IN-US 174-0174
Record Dates: First submitted 2011-11-30; First posted 2011-12-08 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis B Infection; Chronic Infection; Viremia
Keywords: Hepatitis B; Vertical transmission; Pregnancy; Antiviral treatment
MeSH Terms: conditions — Hepatitis B; Persistent Infection; Viremia | interventions — Tenofovir; Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm: HBIG & vaccine for infants (No Intervention): Provide standard of care to mothers and standard immunoprophylaxis to their infants
- TDF treatment arm (Experimental): tenofovir from 30-32 weeks of pregnancy to the week 4 of postpartum for mothers and standard immunoprophylaxis to their infants
  Interventions: Drug: TDF treatment

INTERVENTIONS:
Drug: TDF treatment — About 100 mothers treated with tenofovir from 30-32 weeks of pregnancy to the week 4 of postpartum, then observed to the end of the study at post-partum week 28, paired infants received standard HBV prophylaxis.
  Other Names: Viread, Tenofovir, TDF, Hepatitis B-IgG, Hepatitis B vaccine
  Arms: TDF treatment arm

SUMMARY:
Immunoprophylaxis failure of hepatitis B virus (HBV) leading to vertical transmission remains a concern and has been reported in approximately 8-15% of infants born to hepatitis B e antigen (HBeAg) positive mothers with high levels of HBV DNA. Maternal HBV DNA > 6log10 copies/mL (or >200,000 IU/mL) is the major risk for the mother-to-child transmission. Prior observational studies have shown that antiviral therapy including lamivudine or telbivudine use during late pregnancy can safely reduce the rate of vertical transmission in this special population compared to untreated patients.

Tenofovir Disoproxil (TDF), a pregnancy category B medication, reduces HBV DNA and normalizes serum alanine aminotransferase (ALT) in chronic hepatitis B patients (CHB) with few adverse effects. Two aspects on tenofovir use in pregnancy will be evaluated prospectively in this study:

1. The data on its tolerability and safety in HBeAg+ pregnant women with HBV DNA > 6log10 copies/mL (or > 200,000 IU/mL) during late pregnancy and infants.
2. Its efficacy in the reduction of HBV vertical transmission rate.

DETAILED DESCRIPTION:
Eligible mothers will be randomized (1:1) to either TDF-treated group or untreated group with about 100 subjects in each arm. The treatment group will receive TDF starting at week 30-32 of gestation until week 4 postpartum; follow up will continue until post-partum week 28 and infants age of 28 weeks. Untreated group will receive the standard of care with similar follow-up schedule as the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* documented CHB infection with HBsAg positive > 6 months
* HBeAg+ CHB pregnant women
* gestational age between 30-32 weeks
* HBV DNA > 6 log10 copies/mL (or >200,000 IU/mL)
* both mother and father of the child are willing to consent for the study

Major Exclusion Criteria:

* co-infection with hepatitis A, C, D, E, HIV-1 or sexually transmitted disease (STD)
* decompensated liver disease or significant co-morbidity
* history of abortion, or diagnosis of fetal defect, or congenital malformation in prior pregnancy
* antiviral used within six months prior to this pregnancy, or history of renal or tubular function impairment due to adefovir.
* requirement for other medication during pregnancy to manage other chronic disease(s) or concurrent treatment with immune-modulators, cytotoxic drugs, or steroids
* the biological father of the child had CHB
* clinical signs of threatened miscarriage in early pregnancy
* evidence of hepatocellular carcinoma
* maternal alanine aminotransferase (ALT) > or = 5 x upper limit of normal (U/mL), or Total Bilirubin > or = 2, or glomerular filtration rate (GFR) < 100, or Albumin < 25 g/L
* evidence of fetal deformity by ultrasound examination
* patient is participating other clinical study

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2014-04-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Measure the number of infants who have HBV infection at the age of 28 weeks | From the date of birth to age of 28 weeks
Assessment of the safety and tolerability of TDF, measure the number of participants and paired infants with adverse events | From the date of randomization until 28 weeks of postpartum.

SECONDARY OUTCOMES:
Measure maternal HBV DNA reduction during the study period when compared to the baseline | From the date of radomization to the time of delivery (upto 12 weeks from the radomization)
Measure maternal HBV DNA reduction during the study period when compared to the baseline | From the date of radomization to the time of delivery (about 8 - 10 weeks from the radomization)
percentage of mothers with sero-negativity or sero-conversion of HBsAg and/or HBeAg in each group for comparison | From the date of randomization until 28 weeks of postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Q Pan, MD, Study Chair — Leading Principle Investigator, Division of Gastroenterology and Hepatology, NYU Langone Medical Center, New York; Zhongping Duan, MD, Study Director — Capital Medical University; Shuqin Zhang, MD, Principal Investigator — Hepatobiliary Disease Hospital of Jilin Province, Jilin, China; Erhei Dai, MD, Principal Investigator — The Fifth Hospital of Shijiazhuang, Shijiazhuang, Hebei, China; Guorong Han, MD, Principal Investigator — The Second Affiliated Hospital of the Southeast University, Nanjing, China; Huaihong Zhang, MD, Principal Investigator — Nanyang Central Hospital, Nanyang, Henan, China; Yuming Wang, MD, Principal Investigator — Southwest Hospital, Chongqing, Chongqing, China
Locations (5):
- China (5):
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - The Fifth Hospital of Shijiazhuang, Shijiazhuang, Hebei
  - Nanyang Central Hospital, Nanyang, Henan
  - The Second Affiliated Hospital of the Southeast University, Nanjing, Jiangsu
  - Hepatobiliary Disease Hospital of Jilin Province, Changchun, Jilin

REFERENCES:
- [Derived] Pan CQ, Dai E, Duan Z, Han G, Zhao W, Wang Y, Zhang H, Zhu B, Jiang H, Zhang S, Zhang X, Zou H, Chen X, Chen Y. Long-term safety of infants from mothers with chronic hepatitis B treated with tenofovir disoproxil in China. Gut. 2022 Apr;71(4):798-806. doi: 10.1136/gutjnl-2020-322719. Epub 2021 Mar 31. PMID 33789963
- [Derived] Pan CQ, Duan Z, Dai E, Zhang S, Han G, Wang Y, Zhang H, Zou H, Zhu B, Zhao W, Jiang H; China Study Group for the Mother-to-Child Transmission of Hepatitis B. Tenofovir to Prevent Hepatitis B Transmission in Mothers with High Viral Load. N Engl J Med. 2016 Jun 16;374(24):2324-34. doi: 10.1056/NEJMoa1508660. PMID 27305192